CLINICAL TRIAL: NCT03562923
Title: A Randomized Single Blind Placebo-Controlled Multi-Center Study Comparing Combination Therapy With Fluticasone Propionate 100 mcg and Salmeterol 50 mcg Inhalation Powder to Combination Therapy With ADVAIR DISKUS® 100/50 (Fluticasone Propionate 100 mcg and Salmeterol 50 mcg Inhalation Powder) in Treatment of Subjects With Asthma
Brief Title: A Study to Compare Fluticasone Propionate 100mcg/Salmeterol 50 mcg Inhalation Powder to Advair Discus 100/50
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amneal Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI-FSX-001
Record Dates: First submitted 2018-05-25; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Test Product (Experimental): Test Product, 100/50 mcg, 2 x daily
  Interventions: Drug: Test Product
- Reference Product (Active Comparator): Reference Product, 100/50 mcg, 2 x daily
  Interventions: Drug: Reference Product
- Placebo (Placebo Comparator): Placebo Product 2 x daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Test Product — Fluticasone Propionate 100 mcg and Salmeterol 50 mcg Inhalation Powder
  Arms: Test Product
Drug: Reference Product — ADVAIR DISKUS® 100/50 (Fluticasone Propionate 100 mcg and Salmeterol 50 mcg Inhalation Powder)
  Other Names: ADVAIR DISKUS
  Arms: Reference Product
Drug: Placebo — Placebo Product
  Arms: Placebo

SUMMARY:
To compare the efficacy and safety profiles of Fluticasone Propionate 100 mcg and Salmeterol 50 mcg Inhalation Powder (test product) and ADVAIR DISKUS (fluticasone propionate 100 mcg and salmeterol 50 mcg inhalation powder) (reference product) and to show that the efficacy of the 2 active products is superior to that of placebo in the treatment of subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects (≥ 12 years of age) of non-child bearing potential or of child bearing potential committing to consistent and correct use of an acceptable method of birth control.
* Diagnosed with asthma as defined by the National Asthma Education and Prevention Program (NAEPP) at least 12 weeks prior to screening.
* Pre-bronchodilator FEV1 of ≥40% and ≤85% of the predicted value during the screening visit and on the first day of treatment.
* Currently non-smoking; had not used tobacco products (i.e., cigarettes, cigars, pipe tobacco) within the past year, and had ≤ 10 pack-years of historical use.
* ≥15% reversibility of FEV1 within 30 minutes following 360 mcg of albuterol inhalation (pMDI).
* Able to discontinue their asthma medications (inhaled corticosteroids and long-acting β agonists) during the run-in period and for remainder of the study.
* Able to replace current short-acting β agonists (SABAs) with salbutamol/albuterol inhaler for use as needed for the duration of the study (subjects should be able to withhold all inhaled SABAs for at least 6 hours prior to lung function assessments on study visits).
* Able to continue the following medications without a significant adjustment of dosage, formulation, dosing interval for the duration of the study, and judged able by the investigator to withhold them for the specified minimum time intervals prior to each clinic visit:

  * short-acting forms of theophylline 12 hours
  * twice-a-day controlled-release forms of theophylline 24 hours
  * once-a-day controlled-release forms of theophylline 36 hours
  * Able to discontinue the following medications for the specified minimum time intervals prior to the run-in period and for the remainder of the study:
  * oral corticosteroids 1 month
  * parenteral corticosteroids 1 month
  * oral short-acting β-agonists 12 hours
* Willingness to give their (and in the case of a minor their parent/guardian was able to give) written informed consent to participate in the study.

Exclusion Criteria:

* Life-threatening asthma, defined as a history of asthma episode(s) requiring intubation, and/or associated with hypercapnoea; respiratory arrest or hypoxic seizures, asthma related syncopal episode(s), or hospitalizations within the past year or during the run-in period.
* Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition, historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbated during the study.
* Hypersensitivity to any sympathomimetic drug (e.g., salmeterol or albuterol) or any inhaled, intranasal, or systemic corticosteroid therapy.
* Medication(s) with the potential to affect the course of asthma or to interact with sympathomimetic amines, e.g.:

  * β-blockers
  * oral decongestants
  * benzodiazepines
  * digitalis
  * phenothiazines
  * polycyclic antidepressants
  * Monoamine oxidase inhibitors
* Viral or bacterial, upper or lower respiratory tract infection or sinus or middle ear infection within 4 weeks prior to the screening visit or during the run-in period.
* Factors (e.g., infirmity, disability or geographic location) that the investigator felt would likely limit the patient's compliance with the study protocol or scheduled clinic visits.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1204 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Baseline-adjusted area under the serial FEV1-time curve | 0-12 hours after dosing on day 1
  Baseline-adjusted area under the serial FEV1-time curve calculated from time zero to 12 hours (AUC0-12h) on the first day of treatment.
Baseline-adjusted, pre-dose FEV1 | 4-weeks
  Baseline-adjusted, pre-dose FEV1 on the last day of a 4-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Irshad Haque, Study Director — Amneal Pharmaceuticals, LLC